CLINICAL TRIAL: NCT01389414
Title: Phase II, Open-label, Randomized Clinical Trial of Panitumumab Plus Gemcitabine and Oxaliplatin (GEMOX) Versus GEMOX Alone as First Line Treatment in Advanced Biliary Tract Adenocarcinoma
Brief Title: Panitumumab Plus Gemcitabine and Oxaliplatin (GEMOX)Versus GEMOX Alone to Treat Advanced Biliary Tract Adenocarcinoma
Acronym: Vecti-BIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Massimo Aglietta (Other)
Responsible Party: Sponsor-Investigator, Prof. Massimo Aglietta, Professor, Fondazione del Piemonte per l'Oncologia
Organization: Fondazione del Piemonte per l'Oncologia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-017428-17
Record Dates: First submitted 2011-07-01; First posted 2011-07-08 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Biliary Carcinoma
Keywords: cholangiocarcinoma; biliary; gallbladder; intrahepatic; extrahepatic
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Panitumumab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A- p-Gemox (Experimental): Panitumumab will be administered by intravenous (IV) infusion at a dose of 6 mg/kg once Q2W.
  GEMOX chemotherapy will be administered after the administration of panitumumab once Q2W.
  Gemcitabine 1000mg/sqm will be administered by intravenous infusion as 1-hour infusion on day 1 of each cycle. Oxaliplatin 100mg/sqm will be administered by intravenous infusion as 2-hour infusion on day 2 of each cycle.
  Interventions: Drug: Panitumumab plus GEMOX chemotherapy; Drug: GEMOX chemotherapy
- Arm B-GEMOX (Active Comparator): Gemcitabine 1000mg/sqm will be administered by intravenous infusion as 1-hour infusion on day 1 of each cycle. Oxaliplatin 100mg/sqm will be administered by intravenous infusion as 2-hour infusion on day 2 of each cycle.
  Interventions: Drug: GEMOX chemotherapy

INTERVENTIONS:
Drug: Panitumumab plus GEMOX chemotherapy — panitumumab 6 mg/kg will be administered over 60 minute +/- 15 minutes on day 1 followed by Gemcitabine 1000mg/sqm administered by intravenous infusion as 1-hour infusion on day 1 of each cycle. Oxaliplatin 100mg/sqm will be administered by intravenous infusion as 2-hour infusion on day 2 of each cycle.
  Other Names: panitumumab: Vectibix; Gemcitabine; Oxaliplatin
  Arms: Arm A- p-Gemox
Drug: GEMOX chemotherapy — Gemcitabine 1000mg/sqm will be administered by intravenous infusion as 1-hour infusion on day 1 of each cycle. Oxaliplatin 100mg/sqm will be administered by intravenous infusion as 2-hour infusion on day 2 of each cycle.
  Other Names: Gemcitabine; Oxaliplatin

SUMMARY:
This is a multi-centre phase II, open-label, randomized (1:1), parallel-arm, study of panitumumab in combination with chemotherapy (P-GEMOX) versus chemotherapy alone (GEMOX). Eligible subjects will be enrolled and randomized to receive first-line combination therapy consisting of panitumumab and GEMOX (experimental arm) or GEMOX alone (control arm).The ame of the Stuy is to evaluate the clinical activity of the P-GEMOX (Panitumumab and GEMOX) combination compared to GEMOX alone in patients with previously untreated surgically unresectable or metastatic biliary tract carcinoma (KRAS wild-type)and To evaluate the safety profile of the P-GEMOX combination; to assess the objective response rate; to assess overall survival; to study the correlation between biomarkers with activity and efficacy.

DETAILED DESCRIPTION:
Study Phase: Phase II, Open-label, Randomized

Indication: First line treatment in advanced intrahepatic cholangiocarcinoma and extrahepatic biliary adenocarcinoma including gallbladder.

Primary Objective: To evaluate the clinical activity of the Panitumumab and GEMOX (P-GEMOX) combination compared to GEMOX alone in patients with previously untreated surgically unresectable or metastatic biliary tract carcinoma (KRAS wild-type).

Secondary Objectives: To evaluate the safety profile of the P-GEMOX combination; to assess the objective response rate; to assess overall survival; to study the correlation between biomarkers with activity and efficacy.

Study Design: Multi-centre phase II, open-label, randomized (1:1), parallel-arm, study of panitumumab in combination with chemotherapy (P-GEMOX) versus chemotherapy alone (GEMOX). Eligible subjects will be enrolled and randomized to receive first-line combination therapy consisting of panitumumab and GEMOX (experimental arm) or GEMOX alone (control arm).

Prior to study entry and in order to confirm eligibility, the investigator will review relevant clinical documents including existing radiological images to ensure the subject has previously untreated, unresectable biliary tract adenocarcinoma including gallbladder.

Treatment assignment will be done centrally via an Interactive Voice Response System (IVRS), using a permuted-block randomization stratified according to ECOG performance status (PS) (0 or 1 vs 2), and site of primary tumor (intrahepatic cholangiocarcinoma vs extrahepatic biliary carcinoma including gallbladder).

Panitumumab will be administered by intravenous (IV) infusion at a dose of 6 mg/kg once every two weeks (Q2W).

GEMOX chemotherapy will be administered after the administration of panitumumab once Q2W.

Each patient will be treated for a maximum of 12 cycles until disease progression (PD), unacceptable toxicity, or patient's refusal. Patients in the experimental arm without tumor progression at the end of chemotherapy (12 GEMOX completed or interruption for unacceptable toxicity from chemotherapy) will continue panitumumab 6 mg/kg once Q2W until tumor progression.

Following documentation of progressive disease patients will be followed-up for survival.

Subjects will be evaluated for tumor progression every 8 weeks + 1 week. Tumor response assessment will be performed by the Investigator using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, version 1.1.

Subjects with symptoms suggestive of PD should be evaluated for tumor progression at the time the symptoms occur.

Endpoints:

Primary Endpoint: Progression-free survival (PFS), defined as the time from randomization to evidence of progression (RECIST, vers.1.1), death, or last radiographic assessment in absence of a PFS event.

Secondary Endpoints: Objective response rate (RECIST, vers.1.1); Overall survival; Safety, defined as incidence and severity of adverse events (Aes), significant laboratory changes, changes in vital signs, incidence of concomitant medications, changes from baseline over time in ECOG performance status, incidence of dose adjustments over the treatment period, and incidence of treatment limiting toxicities (TLT).

Exploratory Endpoints:Investigation into potential correlations between the activity of the combination regimen of panitumumab and GEMOX (P-GEMOX) on molecular markers. Depending on the availability of tumor tissue, the biomarkers will be analyzed with the following priority: EGFr expression, nucleotide changes in EGFr and BRAF cancer genes, mutations of other genes involved in the activation of the EGFr pathway; EGFr gene amplification).

Sample Size: Approximately 88 subjects

Investigational Product Dosage and Administration:

Panitumumab will be administered as a 60 minute +/- 15 minutes IV infusion, just prior to administration of chemotherapy, at a dose of 6 mg/kg on day 1 of each cycle. Gemcitabine 1000mg/sqm will be administered by intravenous infusion in accordance with the hospital guidelines for administration of Gemcitabine. Gemcitabine should be reconstituted and administered as 1-hour infusion on day 1 of each cycle. Oxaliplatin 100mg/sqm will be administered by intravenous infusion in accordance with the hospital guidelines for administration of Oxaliplatin. Oxaliplatin should be reconstituted and administered as 2-hour infusion on day 2 of each cycle.

Dose Regimen:

Arm A: panitumumab 6 mg/kg will be administered over 60 minute +/- 15 minutes on day 1 followed by Gemcitabine 1000mg/sqm administered by intravenous infusion as 1-hour infusion on day 1 of each cycle. Oxaliplatin 100mg/sqm will be administered by intravenous infusion as 2-hour infusion on day 2 of each cycle.

Arm B: Gemcitabine 1000mg/sqm will be administered by intravenous infusion as 1-hour infusion on day 1 of each cycle. Oxaliplatin 100mg/sqm will be administered by intravenous infusion as 2-hour infusion on day 2 of each cycle.

Statistical Considerations: This phase II design implies a direct, but non-definitive, "screening" comparison of the experimental therapeutic approach against a randomized standard-treatment control arm, within a trial with a moderate sample size.

Assuming an accrual time of 24 months and a follow-up time of 12 months, accounting for a 10% loss to follow-up in both arms, a total sample of 88 patients is expected to yield the necessary numbers of events if the accrual rate is constant.

The log-rank analysis will be stratified by ECOG PS (0 to 1 vs 2), and site of primary tumor (ie. intrahepatic cholangiocarcinoma vs extrahepatic biliary tract carcinoma including gallbladder).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented surgically unresectable or metastatic biliary tract adenocarcinoma (KRAS wild-type) including gallbladder either at diagnosis or relapsing after surgery.
* Documented KRAS status either on primary tumor or metastasis. KRAS testing will be performed as per center procedure (no centralized analysis is required).
* Availability of a tumor biopsy for the study of tumor biomarkers potentially involved in the response/resistance mechanisms.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* Estimated life expectancy of at least 3 months.
* Adequate bone marrow, hepatic, and renal function determined within 2 weeks prior to starting therapy, defined as:

  * absolute neutrophil count (ANC) ≥ 1.5 x 10E9 cells/L
  * platelet count ≥ 100 x 10E9 cells/L
  * total hemoglobin > 9.0 g/dL
  * total bilirubin < 2.0 x institutional upper limit of normal (ULN)
  * alanine aminotransferase (ALT), aspartate transaminase (AST) < 2.5 x ULN - alkaline phosphatase < 3.0 x ULN
  * creatinine < 1.5 X ULN
  * magnesium ≥ LLN
  * calcium ≥ LLN
* Voluntary, written and dated informed consent.

Exclusion Criteria:

* Any previous chemotherapy or target therapy .
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Coexisting malignancies, except for basal or squamous cell carcinoma of the skin or other solid tumors curatively treated with no evidence of disease for ≥ 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Every 8±1 Weeks until PD
  Progression-free survival (PFS), defined as the time from randomization to evidence of progression (RECIST, vers.1.1), death, or last radiographic assessment in absence of a PFS event.

SECONDARY OUTCOMES:
Objective response rate | Every 8±1 Weeks
  Objective response rate measured by RECIST, vers.1.1
Overall survival | months from randomization to death
  Continuosly verified during the treatment period. After the completion of the treatment to be assessed every 3 months by phone contact.
safety | from the first study drug administration to 28+/-7 days after the last administration
  defined as incidence and severity of adverse events, significant laboratory changes, changes in vital signs, incidence of concomitant medications, changes from baseline over time in ECOG PS, incidence of dose adjustments over the treatment period, and incidence of treatment limiting toxicities (TLT) (Any grade 4 or grade 5 toxicity for any adverse event according to the NCTC, ver. 3).
  Continuosly verified during the treatment period. After the completion of the treatment to be assessed at 28+/-7 days after the last administration.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Aglietta, MD, Principal Investigator — IRCC Candiolo
Locations (12):
- Italy (12):
  - AOU Ospedali Riuniti di Ancona, Ancona, Ancona
  - UO Oncologia Medica Spedali Civili di Brescia, Brescia, Brescia
  - I.R.S.T., Meldola, Meldola
  - San Raffaele Scientific Institute, Milan, Milano
  - Ospedale Niguarda " Ca'-Granda", Milan, Milano
  - Istituto Nazionale per lo studio e la cura dei Tumori-Fondazione Pascale, Napoli, Napoli
  - SC Oncologia Medica Ospedale S.Maria della Misericordia, Perugia, Perugia
  - Centro di Riferimento Oncologico INT di Aviano, Aviano, Pordenone
  - Ircc Candiolo, Candiolo, Torino
  - AOU S.Luigi Gonzaga, Orbassano, Torino
  - A.O.U S.Giovanni Battista, Torino, Torino
  - A.O.U S.Maria della Misericordia, Udine, Udine

REFERENCES:
- [Derived] Leone F, Marino D, Cereda S, Filippi R, Belli C, Spadi R, Nasti G, Montano M, Amatu A, Aprile G, Cagnazzo C, Fasola G, Siena S, Ciuffreda L, Reni M, Aglietta M. Panitumumab in combination with gemcitabine and oxaliplatin does not prolong survival in wild-type KRAS advanced biliary tract cancer: A randomized phase 2 trial (Vecti-BIL study). Cancer. 2016 Feb 15;122(4):574-81. doi: 10.1002/cncr.29778. Epub 2015 Nov 5. PMID 26540314